CLINICAL TRIAL: NCT01772667
Title: Long Term Effects of a 3-week Inpatient Pulmonary Rehabilitation Program in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Long Term Effects of an Inpatient Pulmonary Rehabilitation Program in Patients With Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician of the Department of Pulmology, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Fibrosis2013
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: pulmonary fibrosis; interstitial lung disease; pulmonary rehabilitation; exercise capacity; physical activity; quality of life
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Lung Diseases, Interstitial; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Usual care during the whole study period without pulmonary rehabilitation. The patients will perform their normal daily life.
- Inpatient Rehabilitation (Active Comparator): 3-week inpatient multimodal pulmonary rehabilitation program, including daily exercise training, breathing therapy, medical treatment and psychological support. In the following 3 month, the patients will perform their normal daily life.
  Interventions: Procedure: Inpatient Rehabilitation

INTERVENTIONS:
Procedure: Inpatient Rehabilitation — Rehabilitation program in "Schoen Klinik Berchtesgadener Land"
  Arms: Inpatient Rehabilitation

SUMMARY:
There is evidence that an inpatient pulmonary rehabilitation of 3 weeks improves exercise capacity and quality of life in patients with idiopathic pulmonary fibrosis. However, there are no data available regarding long-term effects of this multimodal program. The aim of this study is to investigate the long-term impact of a rehabilitation program 3 month after finishing on exercise capacity and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* want to start a rehabilitation program in "Schoen Klinik Berchtesgadener Land"
* patients with idiopathic pulmonary fibrosis (vital capacity > 50% pred.)

Exclusion Criteria:

* exacerbation in the last 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Delta of 6-minute walking distance from 1 week pre rehabilitation to 3 month post rehabilitation | 1 week before rehabilitation to 3 month after finishing rehabilitation

SECONDARY OUTCOMES:
Delta of physical activity level from 1 week pre rehabilitation to 3 month post rehabilitation | 1 week before rehabilitation to 3 month after finishing rehabilitation
Delta of SF36-score (questionnaire to measure quality of life) from 1 week pre to 3 month post rehabilitation | 1 week before rehabilitation to 3 month after finishing rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, MD, Study Director — Head physician in the department of pulmology
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany